CLINICAL TRIAL: NCT04341428
Title: A Multi-center, Double-Blind, Randomized, Active-controlled, Parallel-group, Phase III Clinical Trial to Evaluate the Efficacy and Safety of DWP14012 as Maintenance Therapy in Patients With Healed Erosive Esophagitis
Brief Title: Study to Evaluate the Efficacy and Safety of DWP14012 on Maintaining Healing in Subjects With Healed Erosive Esophagitis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DW_DWP14012303
Record Dates: First submitted 2020-04-09; First posted 2020-04-10 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-07

CONDITIONS: Healed Erosive Esophagitis
MeSH Terms: interventions — fexuprazan; Lansoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DWP14012 20mg (Experimental): Orally, once daily
  Interventions: Drug: DWP14012 20 mg; Drug: Lansoprazole 15 mg Placebo
- Lansoprazole 15mg (Active Comparator): Orally, once daily
  Interventions: Drug: DWP14012 20 mg placebo; Drug: Lansoprazole 15 mg

INTERVENTIONS:
Drug: DWP14012 20 mg — DWP14012 20 mg, tablet, orally, once daily for up to 24 weeks
  Arms: DWP14012 20mg
Drug: DWP14012 20 mg placebo — DWP14012 20 mg placebo-matching tablet, orally, once daily for up to 24 weeks
  Arms: Lansoprazole 15mg
Drug: Lansoprazole 15 mg — Lansoprazole 15 mg capsule, orally, once daily for up to 24 weeks
  Arms: Lansoprazole 15mg
Drug: Lansoprazole 15 mg Placebo — Lansoprazole 15 mg Placebo capsule, orally, once daily for up to 24 weeks
  Arms: DWP14012 20mg

SUMMARY:
This study aims to demonstrate the noninferiority of DWP14012 to Lansoprazole 15 mg in the maintenance effect of treatment and confirm the safety of DWP14012 in patients with healed erosive esophagitis confirmed on EGD after medication treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 19 to 75 years, at the date the written informed consent form is signed
2. Subjects with erosive esophagitis (LA Grade A-D) confirmed on EGD within 12 weeks from Visit 2 (randomization day)
3. Subjects with healed erosive esophagitis (no mucosal break observed according to LA classification) confirmed on EGD performed within 10 days before Visit 2 (randomization day) after receiving the standard dose of medicinal products of erosive esophagitis (PPI, P-CAB, etc.) for 4 to 8 weeks for the treatment of erosive esophagitis

Exclusion Criteria:

1. Subjects who have Barrett's esophagus (> 3 cm), gastroesophageal varix, esophagostenosis, ulcer stenosis, active peptic ulcer, acute gastrointestinal bleeding, or a malignant tumor upon EGD screening
2. Subjects who have inflammatory bowel disease (Crohn disease, ulcerative colitis, etc.), irritable bowel syndrome (IBS), primary esophageal motility, or pancreatitis.
3. Subjects with history of clinically significant disease of hepatic, renal, nervous, pulmonary, endocrine, hemato-oncologic, cardiovascular or urinary system
4. Subjects who have had a malignant tumor in the last 5 years
5. Subjects who must continue to take non-steroidal anti-inflammatory drugs (aspirin, etc.), antithrombotic drugs, etc. during the study period (A low dose of aspirin [100 mg/day] which has been administered for prophylactic purpose before study entry is allowed)
6. Subjects who cannot stop the existing erosive esophagitis treatment being taken

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 406 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2021-08-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion (%) of subjects with remission maintained on esophagogastroduodenoscopy by Week 24 | at 24 week

SECONDARY OUTCOMES:
Proportion (%) of subjects with remission maintained on esophagogastroduodenoscopy by Week 12 | at 12 week

OTHER OUTCOMES:
GERD-Health related quality life(HRQL) | at Weeks 4, 12, and 24
  Changes from baseline in the total score of GERD-HRQL at Weeks 4, 12, and 24(The total score could range from 0 to 50 and lower score was evaluated as higher quality of life)
Assessment on symptoms | Weeks 4, 12, and 24
  Proportions of subjects without the major symptoms (heartburn and/or acid regurgitation) at Weeks 4, 12, and 24

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul, South Korea